CLINICAL TRIAL: NCT06494553
Title: Effect of Cervical Stabilization Exercises on Proprioception and Hand Grip Strength in Sedentary Office Workers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shimaa sayed attia, Doctor of Physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSE in SOW
Record Dates: First submitted 2024-06-25; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Cervical Pain
MeSH Terms: conditions — Neck Pain | interventions — Ultrasonic Therapy

STUDY DESIGN:
Intervention Model Description: Pre and post randomized control trial design will be used in this study
Masking Description: Simple randomization was done as the following the name of each subject was written on a paper folding it and putting it in a box; finally papers were picked and assigned to two groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Received traditional treatment program in the form of US, IR and therapeutic exercise program that consisted of Stretching exercises included the following: 1) stretching pectoralis muscle, placing both hands on the occipital area and pulling the elbows back up, and performing arm abduction and external rotation. 2) Stretching the cervical extensors, placing both hands on the occipital area in a sitting position followed by a flexed neck posture with the head down to stretch the cervical extensors .
  Interventions: Device: Ultrasound therapy; Other: traditional treatment program; Device: Infrared therapy
- cervical stabilization exercises group (Experimental): Received cervical stabilization exercises (included the following: Chin tuck, cervical extension, Shoulder shrugs, Shoulder rolls, Scapular retraction) was given in 3 sets with 10 repetitions for 24 sessions (3 sessions per week for 8 weeks) plus traditional treatment program in the form of US, IR and therapeutic exercise program that consisted of Stretching exercises included the following: 1) stretching pectoralis muscle, placing both hands on the occipital area and pulling the elbows back up, and performing arm abduction and external rotation. 2) Stretching the cervical extensors, placing both hands on the occipital area in a sitting position followed by a flexed neck posture with the head down to stretch the cervical extensors.
  Interventions: Other: cervical stabilization exercises; Device: Ultrasound therapy; Other: traditional treatment program; Device: Infrared therapy

INTERVENTIONS:
Other: cervical stabilization exercises — Neck stabilization exercises included the following: Chin tuck, cervical extension, Shoulder shrugs, Shoulder rolls, Scapular retraction
  Arms: cervical stabilization exercises group
Device: Ultrasound therapy — The Chattanooga Intelect ultrasound made in America. Year of production: 2013. It was clinically proven to provide the best possible treatment outcomes by utilizing a high-quality transducer to ensure maximum ultrasound delivery to the treatment area. The output is a clean, culminated beam with the lowest available beam non-uniformity ratio
Other: traditional treatment program — US, IR and therapeutic exercise program that consisted of Stretching exercises included the following: 1) stretching pectoralis muscle, placing both hands on the occipital area and pulling the elbows back up, and performing arm abduction and external rotation. 2) Stretching the cervical extensors, placing both hands on the occipital area in a sitting position followed by a flexed neck posture with the head down to stretch the cervical extensors.
Device: Infrared therapy — Infrared therapy is a non-invasive treatment modality that uses infrared light to promote healing, reduce pain, and improve circulation. It involves the application of infrared light, which penetrates deep into the tissues, providing therapeutic benefits.

SUMMARY:
The purpose of the study is to evaluate the effect of cervical stabilization exercises on pain intensity level, cervical range of motion, proprioception, and handgrip strength in sedentary office workers.

DETAILED DESCRIPTION:
In recent years, the number of sedentary office workers (SOWs) who work in a seated position for prolonged periods has increased with the development of the information technology industry. SOWs are forced to sit for long periods because of the nature of their work. Changes in physical functions that occur due to rounded shoulders can cause one or more abnormal conditions in a complex structure consisting of the head, neck, and shoulders.

Neck pain is a common condition and one of the leading causes of disability worldwide. Although neck pain can be attributed to traumatic (such as whiplash-associated) disorders, metabolic, neoplastic, inflammatory, or infectious diseases, most neck pain has no discernable cause and is considered idiopathic. Current studies have indicated that one of the main problems in patients with neck pain is cervical proprioception impairment, which leads to cervical sensorimotor control disturbances.

The cervical sensorimotor control disturbances secondary to neck pain are considered a protective response to limit further stimulation of the painful tissue. Such disturbances may, in the long- run, further cause tissue damage, aggravate pain through peripheral and central nervous system sensitization, and promote dysfunctional motion patterns. Body posture can affect the proprioception function of the neck.

There is a significant positive association between prolonged sitting at work and neck pain, implying that there is an increased risk of neck pain for people who are working almost all day in a sitting position (more than 95% of the working time).

Working for at least 20 hours a week. Working for at least 1 year in their current job. To improve posture, many physical therapy methods can be used.

A back extensor strengthening exercises that included the following: at a sitting position: 1) shoulder elevation, 2) shoulder horizontal abduction, and 3) shoulder extension; at a standing position: 4) push up and 5) one arm and the opposite leg lift.

Stretching exercises included the following: 1) stretching pectoralis muscle, placing both hands on the occipital area and pulling the elbows back up, and performing arm abduction and external rotation. 2) Stretching the cervical extensors, placing both hands on the occipital area in a sitting position followed by a flexed neck posture with the head down to stretch the cervical extensors.

Neck stabilization exercises included the following: Chin tuck, cervical extension, Shoulder shrugs, Shoulder rolls, Scapular retraction.

Advises: subjects will be educated to assume good posture and alignment during sitting and standing activities such as: Sitting upright in a chair and not leaning forward, Using pillows behind the lower back, Sitting on a chair with head and arm support.

These programs were selected from programs commonly used in previous studies.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 25 and 35 years.
* Both male and female patients were included.
* Informed consent was obtained from all participants.
* Subjects with cervical pain lasting for more than 3 months (chronic pain).
* Cooperative patients who were able to follow instructions for assessment procedures.
* body mass index (18.5 - 29.99 Kg/m2).

Exclusion Criteria:

* Unwillingness to participate in the treatment.
* Pre-existing heart or respiratory diseases.
* Acute cervical pain.
* Cervical disc or spondylosis.
* History of any major cervical spine surgery.
* Subjects taking analgesics.
* Any fracture of cervical region.

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
handgrip strength | 2 months
  Handgrip strength is a crucial measure of overall muscle strength and function to assess the functionality of the hand and forearm muscles. This measure is typically obtained using a handgrip dynamometer, a device that quantifies the maximum isometric strength of the hand and forearm muscles.
cervical range of motion | 2 months
  Cervical Range of Motion (CROM) refers to the degree of movement in the neck and cervical spine across different planes of motion. It is an important measure of neck flexibility and function, encompassing movements such as flexion, extension, lateral flexion, and rotation. Assessing CROM is crucial in diagnosing and managing various musculoskeletal and neurological conditions affecting the neck.
  This measure is typically obtained using CROM devices that play a pivotal role in accurately quantifying the range of motion in various planes, including flexion, extension, lateral flexion, and rotation.
cervical pain | 2 months
  Cervical pain, commonly known as neck pain, is a prevalent condition characterized by discomfort, stiffness, or aching in the cervical spine-the region of the spine that comprises the neck. This condition can arise from various causes, ranging from muscle strain to more complex structural issues, and it can significantly impact a person's quality of life, daily activities, and functional capabilities.
  This measure is typically obtained using Alternate Visual Analog Scale in Hausa (VAS-H).
  The VAS-H was used to measure the level of pain experienced by the patients. Patients were asked to rate their pain on a scale of 0-10, with 0 indicating no pain/no interference and 10 indicating the worst possible pain/extreme interference. The alternate VAS-H has been shown to have high validity, increased patient compliance, greater sensitivity, and reduced bias.
cervical proprioception | 2 months
  Cervical proprioception refers to the sensory ability of the neck muscles and joints to perceive their position and movement in space. This sensory feedback is critical for maintaining balance, coordinating head and eye movements, and performing complex motor tasks. Impaired proprioception in the cervical region can contribute to dizziness, balance disorders, and increased risk of injury.
  This measure is typically obtained using CROM devices that play a pivotal role in accurately quantifying the range of motion and proprioception in various planes, including flexion, extension, lateral flexion, and rotation.

REFERENCES:
- [Background] Bernal-Utrera C, Gonzalez-Gerez JJ, Anarte-Lazo E, Rodriguez-Blanco C. Manual therapy versus therapeutic exercise in non-specific chronic neck pain: a randomized controlled trial. Trials. 2020 Jul 28;21(1):682. doi: 10.1186/s13063-020-04610-w. PMID 32723399
- [Background] Reddy RS, Tedla JS, Dixit S, Abohashrh M. Cervical proprioception and its relationship with neck pain intensity in subjects with cervical spondylosis. BMC Musculoskelet Disord. 2019 Oct 15;20(1):447. doi: 10.1186/s12891-019-2846-z. PMID 31615495